CLINICAL TRIAL: NCT02506582
Title: The Effects of Jerusalem Artichoke and Fermented Soybean Powder Mixture Supplementation on Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS_DM
Record Dates: First submitted 2015-05-06; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Prediabetes; Newly Diagnosed Type 2 Diabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental): jerusalem artichoke and fermented soybeans powder mixture supplementation
  Interventions: Dietary Supplement: jerusalem artichoke and fermented soybeans powder mixture
- Placebo group (Placebo Comparator): placebo supplementation
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: jerusalem artichoke and fermented soybeans powder mixture — 40 g jerusalem artichoke and fermented soybean powder mixture
  Arms: Test group
Dietary Supplement: placebo — 40 g powdered rice flour
  Arms: Placebo group

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled study was to determine whether jerusalem artichoke and fermented soybeans powder mixture is effective in the control of blood glucose level in subjects with prediabetes or newly diagnosed type 2 diabetes.

DETAILED DESCRIPTION:
The objective of this clinical study was to evaluate the effect of jerusalem artichoke and fermented soybean powder mixture supplementation on blood glucose. A randomized, double-blinded, placebo-controlled study was conducted on 60 subjects with impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or newly diagnosed type 2 diabetes. The subjects were randomly assigned to either a group ingesting 40 g jerusalem artichoke and fermented soybean powder mixture supplementation daily or a placebo group for 12-week. We assessed fasting and postprandial levels of glucose.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects were with prediabetes (IFG or IGT) or newly diagnosed type 2 DM (T2DM) no taking medicine. IFG was defined as fasting glucose between 100 and 125 mg/dL and IGT was defined as 2-h OGTTs glucose levels 140-199 mg/dL. Newly diagnosed type 2 diabetes was defined as fasting glucose ≥126 mg/dL or 2-h OGTTs level ≥ 200 mg/dL.

Exclusion Criteria:

1. glucose lowering medications or insulin injections;
2. abnormal liver or renal function;
3. chronic stomach and intestines disease;
4. chronic alcoholism;
5. pregnancy or intending to become pregnant during time of study.
6. complications;
7. an occupation that could be dangerous if hypoglycemia should occur.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose level by 2-h oral glucose tolerance tests (OGTTs) | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, PhD, Study Chair — Yonsei University